CLINICAL TRIAL: NCT02244853
Title: Association of Heart Rate With Cardiovascular Disease Prognosis of Patients With Stable Coronary Artery Disease: A CALIBER Study
Brief Title: Heart Rate and Cardiovascular Diseases Prognosis in People With Stable Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor, University College, London
Other Study IDs: 12_153R_IP24; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust); RP-PG-0407-10314 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Stable Angina; Myocardial Infarction; Coronary Heart Disease; Heart Failure; Stroke; Death, Sudden, Cardiac; Peripheral Arterial Disease; Atrial Fibrillation; Bleeding
MeSH Terms: conditions — Angina, Stable; Myocardial Infarction; Coronary Disease; Heart Failure; Stroke; Death, Sudden, Cardiac; Peripheral Arterial Disease; Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Cardiovascular disease research using Linked Bespoke studies and Electronic Records (CALIBER) e-health database was the data resource for this study. CALIBER links patient records from four different data sources: Clinical Practice Research Database (CPRD), MINAP (Myocardial Ischaemia National Audit Project registry) Hospital Episodes Statistics (HES), the Office for National Statistics (ONS).

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* Aged >=30 years at study entry ->=1 year registration prior to the 'index date'

Exclusion Criteria:

* Free from previous atherosclerotic events
* No heart rate measurement after their 'index date' of eligibility to entry the study

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An open cohort of 2,23 million people covering approximately 5% of the UK population was drawn from registrants to 225 GP practices who consented to data linkage.
Sampling Method: Non-Probability Sample
Enrollment: 51703 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Risk of cardiovascular diseases in patients with low and high heart rate and stable coronary artery disease | expected average of 3 years
  Participants were followed until their first cardiovascular or complication event after their studyentry and after at least one previous cardiovascular event. Hazard ratios will be presenting associations between heart rate (analysed as quintiles and as continuous per 10bpm) and 8 different cardiovascular diseases (including mortality outcomes, complications such as bleeding events and composite cerebrovascular and coronary heart disease endpoints).

CONTACTS AND LOCATIONS:
Overall Officials: Harry Hemingway, Professor, Study Director — Farr Institute
Locations (1):
- Farr Institute, University College London, London, United Kingdom